CLINICAL TRIAL: NCT01010347
Title: A Comparison of Casting and Splinting in Pediatric Radial Buckle Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-1088
Record Dates: First submitted 2009-11-04; First posted 2009-11-10 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Distal Radial Buckle Fractures
Keywords: fractures; casting; splinting; pediatrics
MeSH Terms: conditions — Fractures, Bone | interventions — POLR1G protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Splint (Active Comparator): Preformed velcro volar splints are compared to traditional circumferential casting.
  Interventions: Procedure: Volar Splint
- Cast (Placebo Comparator): The circumferential cast is the standard of treatment against which the splint is compared.
  Interventions: Procedure: Cast

INTERVENTIONS:
Procedure: Volar Splint — A velcro volar splint is compared to a circumferential cast for the treatment of distal radial buckle fractures in children. These are to be worn until Pediatric Orthopaedics follows up with the patients at 3 weeks.
  Other Names: Biomed Volar Splint
  Arms: Splint
Procedure: Cast — A velcro volar splint is compared to a circumferential cast for the treatment of distal radial buckle fractures in children. These are to be worn until Pediatric Orthopaedics follows up with the patients at 3 weeks.
  Arms: Cast

SUMMARY:
Background: distal radial buckle fractures are common injuries in children. the ideal immobilization technique is controversial. Few, retrospective studies have been conducted to evaluate bone healing after casting versus splinting. However, the impact of the immobilization technique on daily function and comfort has not been evaluated.

Objective: To compare the impact on daily function, comfort and satisfaction of casting versus splinting in children with distal radial buckle fractures.

Primary Hypothesis: Children with short arm casts to immobilize a distal radial buckle fracture will have a greater reduction in daily activities compared to those immobilized with a volar splint.

Secondary Hypothesis: Children who are immobilized in a short arm cast will have less pain, less patient/parental satisfaction, more adverse effects, fewer follow-up visits, longer emergency department (ED) treatment time. Furthermore, we hypothesize that all fractures will have acceptable alignment/healing at the follow-up orthopaedic clinic evaluation.

DETAILED DESCRIPTION:
Methods: A randomized controlled trial will be conducted in children 2 to 17 years old with a radio graphically confirmed distal radial buckle fracture. Exclusion criteria will include skeletal maturity, previous distal radius fracture, concurrent other fracture(s), osteogenesis imperfecta or other metabolic bone disease. Enrolled subjects will be randomized to receive either a short arm cast or a volar wrist splint. The pediatric emergency department attending physician will be responsible for applying or directly supervising the immobilization technique. All subjects' radiographs will be reviewed by a pediatric orthopaedic surgeon with 1 day to confirm diagnosis and measure fracture angulation. Those subjects with unacceptable angulation will be called and asked to return to the ED or orthopaedic clinic for re-evaluation.

Outcomes Measures: The primary outcome measure will be the Peds QL questionnaire to assess impact on daily function. This will be assessed at baseline in the ED, by phone at 1 day, 3 days and 1 week after the ED visit, and at the orthopaedic clinic follow-up visit 3 weeks after the ED visit. Secondary outcome measures will include questionnaires assessing demographic data (baseline), pain, satisfaction, adverse effects (baseline, immediately after immobilization applied, 1 day, 3days and 1 week after ED visit by phone, and at the 3 week orthopaedic clinic follow-up visit), and ED treatment time (in ED prior to discharge). At the 3 week orthopaedic surgery clinic follow-up visit, an assessment of the integrity of the immobilization technique will be conducted by a cast technician and fracture alignment/healing and range of motion of affected arm will be conducted by the pediatric orthopaedic surgeon who will be blinded to treatment group.

ELIGIBILITY:
Inclusion Criteria:

* 2 - 17 years
* radiographically confirmed distal radial buckle fracture

Exclusion Criteria:

* skeletal maturity
* previous distal radius fracture
* concurrent other fracture
* osteogenesis imperfecta or other metabolic bone disease

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the Peds QL questionnaire to assess impact on daily function. | Patients are followed for 3 weeks after the initial emergency encounter. They complete the PedsQL and answer questions by telephone.

SECONDARY OUTCOMES:
Pain and satisfaction. | Patients and parents are queried via telephone at days 1, 3, and 7 after the initial emergency visit. They are questioned about pain scores and satisfaction with the immobilization device.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Williams, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States